CLINICAL TRIAL: NCT03840551
Title: Definition of a Set of Biomechanical Indices Non-invasively Measurable During Basic Sport Movements Test Analysis Aimed to the Prevention of Primary and Secondary Anterior Cruciate Ligament Injury
Brief Title: Definition of Biomechanical Indices Measurable During Sport Movements for the Prevention of Primary and Secondary ACL Injury
Acronym: BIOS-ACL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Isokinetic (Unknown)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Professor, Istituto Ortopedico Rizzoli
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 28/18
Record Dates: First submitted 2019-02-06; First posted 2019-02-15 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Sport Injury; Anterior Cruciate Ligament Injury; Biomechanical; Lesion
Keywords: injury prevention; biomechanical indices; inertial sensors
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Motion Capture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects (Other): Subjects involved are required to do some specific motor tasks, commonly found in all main sports. Evaluated with inertial sensors (XSENS) and marker-based motion capture (BTS)
  Interventions: Other: Biomechanical analysis with inertial sensors (XSENS) and motion capture (BTS)

INTERVENTIONS:
Other: Biomechanical analysis with inertial sensors (XSENS) and motion capture (BTS) — The kinematics of lower limbs, trunk and upper limbs will be calculated both with inertial sensors (XSENS) and motion capture marker-based system (BTS ). Inertial sensors and markers will be placed on the subjects clothes and on the skin (totally non-invasive) to identify body segments. Then subjects will perform their motor tasks normally. Lately, through the data post-processing, the kinematics evaluated with both the systems will be used to describe how well the task is performed in terms of ACL prevention, through derived biomechanical parameters.

SUMMARY:
The aim of the study is to define a set of quantitative parameters related to articular biomechanics, which will be evaluated during some specific motor tasks. The goal is the prevention of primary and secondary anterior cruciate ligament injury in athletes.

Specifically, the validation of a new comparative methodology of biomechanics analysis will be performed, based on inertial sensors and musculoskeletal models. This way, brief but exhaustive description of functional characteristics of athletes could be created and easily used in ambulatory environment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, men of women, 18 years old minimum and 50 maximum, which read and signed the informed consent

Exclusion Criteria:

* evidence of any kind of musculoskeletal disease or impairment
* evidence of past surgical intervention to either lower or upper limbs
* age out of the inclusion range
* cardiac or pulmonary diseases
* inability to read and sign the informed consent
* inability to perform the motor tasks required

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Lower limbs angles (extracted by inertial sensors/motion capture marker-based analysis): Hip, Knee, Ankle joint angles (all in degrees °) | 10 months
  These quantitative parameters are the output of the inertial sensor and marker-based motion capture dedicated softwares, and will be then post processed and analyzed to find the range of motion, the maximum and the minimum angles for each joint. Every outcome angle is expressed in degrees (°)
  * Hip angles (flexion/extension, ab/adduction and intra/extra rotation) in degrees (°);
  * Knee angles (flexion/extension, varus/valgus and intra/extra rotation) in degrees (°);
  * Ankle angles (flexion/extension, ab/adduction and intra/extra rotation) in degrees (°).
Upper limbs angles (extracted by inertial sensors/motion capture marker-based analysis): Elbow, Wrist and Shoulder joint angles (all in degrees °) | 10 months
  These quantitative parameters are the output of the inertial sensor and marker-based motion capture dedicated softwares, and will be then post processed and analyzed to find the range of motion, the maximum and the minimum angles for each joint, and the interaction with lower limbs joint angles. Every outcome angle is expressed in degrees (°)
  * Elbow angles (flexion/extension, intra/extra rotation) in degrees (°);
  * Wrist angles (flexion/extension) in degrees (°);
  * Shoulder angles (flexion/extension, ab/adduction) in degrees (°).
Trunk angles (extracted by inertial sensors/motion capture marker-based analysis): Trunk sway and Trunk tilt (all in degrees °) | 10 months
  These quantitative parameters are the output of the inertial sensor and marker-based motion capture dedicated softwares, and will be then post processed and analyzed to find the range of motion, the maximum and the minimum angles for each joint, and the interaction with lower limbs joint angles. Every outcome angle is expressed in degrees (°)
  * Trunk sway in degrees (°) ;
  * Trunk tilt in degrees (°) .
Trunk velocity (in m/s) extracted by inertial sensors/motion capture marker-based analysis | 10 months
  Trunk velocity in all 3 directions (x,y,z). Expressed in m/s
Trunk acceleration (in m/s^2) extracted by inertial sensors/motion capture marker-based analysis | 10 months
  Trunk Acceleration in all 3 directions (x,y,z). Expressed in m/s^2

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Mr Zaffagnini, Professor, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided